CLINICAL TRIAL: NCT03635697
Title: The Effect of an Auditory Mindfulness Intervention During NST Appointments on Depression and Anxiety in Pregnant Women
Brief Title: Mindfulness in Pregnancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 and guideline changed
Sponsor: UConn Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-226-1
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Depression; Mindfulness
Keywords: Pregnancy; Mindfulness; Anxiety; Depression; NST; Non-stress test
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Intervention Group (Experimental): Participants in this group will listen to a short mindfulness audio clip during 6 of their NST appointments.
  Interventions: Behavioral: Mindfulness Auditory Intervention
- Control Group (No Intervention): Participants in this group will have the regular standard of care for their NST appointments.

INTERVENTIONS:
Behavioral: Mindfulness Auditory Intervention — This intervention is a short audio clip that focuses on the practices and principles of mindfulness. The goal of mindfulness is to bring awareness to a person's physical body as well as their thoughts and feelings.
  Arms: Mindfulness Intervention Group

SUMMARY:
This study aims to determine if a short audio clip about mindfulness implemented during NST appointments can lower pregnant women's levels of anxiety and depression. Subjects will be placed into either the intervention group or a control group. The intervention group will be asked to listen to a short audio clip on mindfulness during their NST appointments, and the control group will receive the standard of care during NST appointments. Subjects will be asked to take two surveys about anxiety and depression three times throughout the study: before the intervention, after the intervention, and 6 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English as primary language
* less than 36 weeks gestational age
* at least 28 weeks gestational age

Exclusion Criteria:

* Use of psychoactive medications
* Any psychiatric diagnosis with dissociative, hallucinatory, and/or delusional features
* History of suicide attempt or current suicidal ideations
* Uncontrolled substance abuse in the last 6 months
* Patients with hearing loss
* More than three no-shows to NST appointments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory Score | Over the course of 6 intervention sessions, followed by 6 weeks postpartum
  We are looking for the members of our intervention group to see a change in their scores on the Beck Anxiety Inventory after completing 6 sessions of listening to a mindfulness clip. We expect to see this score change after the full-course of the intervention is complete. We also hope to see this change in score persist at the 6-week postpartum visit. This scale aims to measure anxiety symptoms, and total scores range from 0-36. Lower scores indicate lower levels of anxiety symptoms, and thus a better outcome.
Edinburgh Postnatal Depression Scale Score | Over the course of 6 intervention sessions, followed by 6 weeks postpartum
  We are looking for the members of our intervention group to see a change in their scores on the Edinburgh Postnatal Depression Scale after completing 6 sessions of listening to a mindfulness clip. We expect to see this score change after the intervention is complete. We also hope to see this change in score persist at the 6-week postpartum visit. This scale aims to measure depressive symptoms, and total scores range from 0-30. Lower scores indicate lower levels of depressive symptoms, and thus a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Morosky, MD, Principal Investigator — UConn Health
Locations (1):
- UConn Health / John Dempsey Hospital, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No